CLINICAL TRIAL: NCT05833165
Title: Feasibility of Integrating Homeopathic Approach in a Comprehensive Cancer Center
Status: Recruiting | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, MOSHE FRENKEL MD, Principal Investigator, Rambam Health Care Campus
Other Study IDs: RMB-0194-22
Record Dates: First submitted 2023-04-03; First posted 2023-04-27 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Quality of Life; Complementary Medicine; Integrative Medicine
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Feasibility of a supportive approach: Evaluating a feasibility of an approach
  Interventions: Behavioral: Feasibility of a supportive approach

INTERVENTIONS:
Behavioral: Feasibility of a supportive approach — Evaluating reasons for patients to use the approach

SUMMARY:
Supportive and palliative care play an important role in cancer treatment, and when introduced early can improve quality of life and may even increase median survival rates, as shown in patients with advanced lung cancer. Complementary and integrative medicine (CIM) is a popular supportive approach among oncology patients and is on the rise worldwide. In many countries, homeopathy is being one the CIM methods integrated with a general sense that this treatment is beneficial to the well-being and quality of life (QoL) of cancer patients. In this observational study we will evaluate the feasibility of integrating homeopathic approach in patients attending the complementary and integrative oncology service at the division of oncology in Rambam Health Campus in Haifa, Israel, a major referral comprehensive cancer center.

This observational study will evaluate three main ingredients of acceptance:

* Obtaining the reasons that patients willing to integrate this supportive approach
* Patient acceptance of this supportive approach as well as compliance with the homeopathic approach
* Obtaining retrospective subjective information from the patients through validated quality of life questionnaires. (MYCaW, Distress Thermometer, and ESAS-R) Measures which are used routinely in integrative oncology encounters.

DETAILED DESCRIPTION:
Supportive and palliative care play an important role in cancer treatment, and when introduced early can improve quality of life and may even increase median survival rates, as shown in patients with advanced lung cancer.

Complementary and integrative medicine (CIM) is a popular supportive approach among oncology patients and is on the rise worldwide. As a response to this demand, there is an understanding that these approaches need to be integrated in cancer care. In 90% of large comprehensive cancer centers in the US and in many others in Europe and elsewhere, complementary and integrative medicine is being integrated into supportive patient care.

In Israel similar trend is observed and 8 integrative oncology services has been established around the country in the majority of oncology centers. Homeopathy is one of the CIM modalities utilized by patients with cancer. It is widely practiced worldwide, especially in Europe, Asia, and Latin America.

In the United States, during the 1990s, sales of homeopathic medicines grew at an annual rate of 20-25%, and in the 2015 US National health statistics report, homeopathy was mentioned as used by over 5 million people.

This modality involves detailed interview that emphasizes the unique characteristics of symptoms experienced by patients followed by utilizing highly diluted substances. Dilutions that are above 12c (dilution of 10-24 actually do not have the original substance), which are commonly used in homeopathy, reflect that the original material is not in this remedy. As a result of this understanding this complementary therapy remains one of the debated modalities in CIM.

Some mention that patients seek that method of care due to the fact that this approach emphasizes empathic listening to patients' concerns and worries, and the effect of the actual remedy, due to its high dilution, reflect a placebo response.

On the other hand, some clinical studies reveal that the use of homeopathy in cancer care, as a supportive approach, reflects clinical benefit that is not attributed to placebo, without risk of side effects or interactions with the conventional oncology approach.

In one prospective observational study done in Germany with cancer patients in two differently treated cohorts: one cohort with patients under complementary homeopathic treatment (n = 259), and one cohort with conventionally treated cancer patients (n = 380). It was observed that an improvement in quality of life was observed in patients taking the addition of homeopathic treatment, as well as a tendency of fatigue symptoms to decrease in cancer patients under complementary homeopathic treatment.

Another recent descriptive study that was conducted in France in three oncology centers in one city. Researchers observed that homeopathy was used in 30% of the cancer patients. (n=633) The homeopathy was used as an additional supportive measure. Fatigue was one of the leading symptoms that improved in 80% of the patients that homeopathy was added to their care.

An Israeli study evaluated the adherence to homeopathic treatment among cancer patients who received a CIM consultation (n=124). The authors found that homeopathy treatment was feasible, with two-thirds of patients acquiring and self-administering the remedies as prescribed. Fatigue was one of the main symptoms that patients felt that improved with the addition of homeopathy.

In another prospective, randomized, placebo-controlled, double-blind, three-arm, multicenter, phase III study at the University of Vienna, researchers evaluated the possible effects of additive homeopathic treatment compared with placebo in 150 patients with stage IV Non-Small Cell Lung Cancer (NSCLC). Researchers found that there was a significant improvement of quality of life measures in the additive homeopathy group when compared with placebo after 9 and 18 weeks of homeopathic treatment. In addition, median survival time was significantly longer in the homeopathy group (435 days) versus placebo (257 days; p = .010) as well as, versus control (228 days; p < .001).

Homeopathy is considered safe and without adverse effects, neither direct (i.e., toxic effects) nor indirect (i.e., interactions with conventional anticancer agents).

In this study, patients affected by cancer that attend the oncology department in Rambam Health Campus, and wish to utilize the CIM service, will be offered this option of care.

The aim of the present study is therefore to evaluate the feasibility of the process of integrating homeopathy as a potential treatment option for symptom control and improvement in quality of life in cancer patients, in a comprehensive cancer center.

This observational study will evaluate three main ingredients:

* Obtaining main concerns of patients that agree to utilize this method
* Patient acceptance of this supportive approach that will be reflected in obtaining and self-administering the remedies as prescribed.
* Obtaining retrospective subjective information from the patients through validated quality of life questionnaires. (MYCaW, Distress Thermometer, and ESAS-R) Measures which are used routinely in integrative oncology encounters, at the initial evaluation, and during follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* • 18 years of age or older

  * Ability to read, write, and understand the Hebrew language
  * Patients treated at the Division of Oncology in Rambam Health Campus.
  * Performance status of ECOG 0-2.
  * Consent to participate in the study.

Exclusion Criteria:

* • Inability to understand the intent of the study and follow the instructions

  * Diagnosis of active psychosis, altered mental state or severe cognitive impairment confirmed by the patient's attending physician.
  * Frailty, ECOG worse than 2, or other unstable medical conditions as confirmed by the patient's attending physician including acute illness, fever, unclear rash or medical conditions that would preclude participation in an interview session lasting 15-30 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that elect to use complementary and integrative medicine during cancer care and make a choice to use homeopathy as part of this use
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a supportive approach | 6-12 weeks
  Questionnaire
Quality of life- Level of Distress | 6-12 weeks
  Distress thermometer

CONTACTS AND LOCATIONS:
Overall Officials: Maria Suleymanov, RN, Study Director — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Theunissen I, Bagot JL. Supportive cancer care: is integrative oncology the future? Curr Opin Oncol. 2024 Jul 1;36(4):248-252. doi: 10.1097/CCO.0000000000001027. Epub 2024 Feb 23. PMID 38842016
- [Background] Frenkel M. Is There a Role for Homeopathy in Cancer Care? Questions and Challenges. Curr Oncol Rep. 2015 Sep;17(9):43. doi: 10.1007/s11912-015-0467-8. PMID 26210222
- [Background] Frass M, Lechleitner P, Grundling C, Pirker C, Grasmuk-Siegl E, Domayer J, Hochmair M, Gaertner K, Duscheck C, Muchitsch I, Marosi C, Schumacher M, Zochbauer-Muller S, Manchanda RK, Schrott A, Burghuber O. Homeopathic Treatment as an Add-On Therapy May Improve Quality of Life and Prolong Survival in Patients with Non-Small Cell Lung Cancer: A Prospective, Randomized, Placebo-Controlled, Double-Blind, Three-Arm, Multicenter Study. Oncologist. 2020 Dec;25(12):e1930-e1955. doi: 10.1002/onco.13548. Epub 2020 Nov 7. PMID 33010094
- [Background] Dolev T, Ben-David M, Shahadi I, Freed Y, Zubedat S, Aga-Mizrachi S, Brand Z, Galper S, Jacobson G, Avital A. Attention Dysregulation in Breast Cancer Patients Following a Complementary Alternative Treatment Routine: A Double-Blind Randomized Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211019470. doi: 10.1177/15347354211019470. PMID 34027702
- [Background] Samuels N, Freed Y, Weitzen R, Ben-David M, Maimon Y, Eliyahu U, Berger R. Feasibility of Homeopathic Treatment for Symptom Reduction in an Integrative Oncology Service. Integr Cancer Ther. 2018 Jun;17(2):486-492. doi: 10.1177/1534735417736133. Epub 2017 Nov 2. PMID 29094627